CLINICAL TRIAL: NCT05933317
Title: A Long-term Follow-up Study of Pulmonary Function Changes Using Phase-resolved Functional Lung MRI in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Tao Ouyang, Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Other Study IDs: 202212301
Record Dates: First submitted 2023-07-05; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Functional lung MRI — Functional lung MRI

SUMMARY:
So far, the number of COVID-19 infections worldwide has exceeded 700 million. Long-term damage to the lungs is a major sequela of COVID infection. Pulmonary function testing is an important means for the evaluation of lung damage. MRI examinations with free breathing and no contrast agent can prevent patients from suffering from ionizing radiation damage caused by multiple CT examinations.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years; Sign the informed consent; Patients diagnosed with COVID-19 by nucleic acid test and survived to be discharged; Complete clinical data during hospitalization.

Exclusion Criteria:

* Patients with bacterial pneumonia; Patients with MRI contraindications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients with COVID-19
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
QDP, VDP | 6 months
  perfusion defect percentage, ventilation defect percentage

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Dr., Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China